CLINICAL TRIAL: NCT07114016
Title: Efficacy of Topical Glucosamine Versus Corticosteroid on Tumor Necrosis Factor -Alpha Induced Apoptosis in Oral Lichen Planus: A Randomized Controlled Clinical Trial With Immunohistochemical Analysis
Brief Title: Efficacy of Topical Glucosamine Versus Corticosteroid in Oral Lichen Planus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Sara Abd El-Halim Galala, Assistant Lecturer of Oral Medicine, Periodontology and Oral Diagnosis, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-REC0787
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Oral Lichen Planus
Keywords: GlcN.H
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Glucosamine; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucosamine (Experimental): (Topical glucosamine hydrochloride 1%) Four times per day for 8 weeks
  Interventions: Drug: Glucosamine Hydrochloride
- Corticosteroids (Active Comparator): Topical steroid (triamcinolone acetonide 0.1 %) four times per day for 8 weeks
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Glucosamine Hydrochloride — GlcN.H is an N-deacetyl amino sugar derived from the complete hydrolysis of chitosan known for its immunoregulatory capacity and anti-inflammatory effects.
  Arms: Glucosamine
Drug: Triamcinolone Acetonide — Topical corticosteroid (triamcinolone acetonide is a synthetic corticosteroid with potent anti-inflammatory, anti-allergic, and immunosuppressive properties which is used commonly in topical formulations)
  Arms: Corticosteroids

SUMMARY:
Glucosamine (GlcN) is an N-deacetyl amino sugar derived from the complete hydrolysis of chitosan. It is classified as a nutraceutical and it is used mainly orally for the therapy of osteoarthritis since GlcN has immunoregulatory capacity and anti-inflammatory effects. Given the Oral lichen planus (OLP) T-cell-mediated pathogenesis; this drug seems to be a promising therapeutic option. The investigators compared the clinical efficacy of topical glucosamine to topical corticosteroid in the treatment of symptomatic OLP and investigated the effect of these two treatment modalities on the expression of tumor necrosis factor-alpha (TNF-α) in oral lichen planus lesions

DETAILED DESCRIPTION:
Thirty-six patients with erosive or atrophic OLP were randomly assigned into Two equal groups to receive topical GlcN (glucosamine hydrochloride 1%) 4 times/day for 8 weeks (Group I) and topical steroid (triamcinolone acetonide 0.1 %) 4 times / day for 8 weeks (Group II). All patients were followed up for another 4 weeks (treatment free observational period). Photographs of the most severe lesion were taken (Marker lesion) in each patient and analyzed for total surface area (TSA), total ulcerative area (TUA), total atrophic area (TAA), and total papular area (TPA), patients were also assessed using clinical scores (CS) and visual analogue scale (VAS). Pre-treatment and post-treatment specimens were immunohistochemically analyzed to detect expression of TNF-α.

ELIGIBILITY:
Inclusion Criteria:

* Clinically proven painful bullous/erosive or atrophic forms of OLP
* Histopathologically proven bullous/erosive or atrophic forms of OLP

Exclusion Criteria:

* Lichenoid lesions.
* Presence of systemic conditions
* Smoking.
* Hypersensitivity or severe adverse effects to the treatment drugs or to any ingredient of their preparation as mentioned in medical history.
* Pregnancy or breast-feeding.
* Presence of skin lesions.
* History of previous treatments potentially effective on OLP.
* Loss of pliability or flexibility in the tissues involved by the oral lesions of lichen planus.
* Histological signs of epithelial dysplasia or lichenoid lesions within the biopsied sites.
* Refusing to participate in the study.
* Vulnerable groups

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Clinical score (CS) | Change from Baseline at 12 weeks
  "0" represented no lesion/normal mucosa; "1" mild white striae/no erythematous area, "2"white striae with atrophic area less than 1 cm², "3" white striae with atrophic area more than 1 cm², "4" white striae with erosive area less than 1 cm², and "5" white striae with erosive area more than 1 cm²

SECONDARY OUTCOMES:
TNF-α | Change from baseline at 8 weeks
  TNF-α is a highly pleiotropic multifunctional cytokine. It plays a prominent role in host defense and immune responses to infection, influences remodeling of tissue, angiogenesis stimulation and takes part in regulation of cell proliferation and differentiation. It has been known as an important mediator of cancer

OTHER OUTCOMES:
Visual Analogue Scale (VAS) | Change from Baseline at 12 weeks
  Patients ranked the severity of pain on 10-cm visual analogue scale from (0 to10) where "0" represented no pain to "10" represented the worst pain
TSA | Change from Baseline at 12 weeks
  Total area of the marker lesion (mm2)
TUA | Change from Baseline at 12 weeks
  Surface area of ulcer in marker lesion (mm2)
TAA | Change from Baseline at 12 weeks
  Surface area of atrophic areas in marker lesion (mm2)
TPA | Change from Baseline at 12 weeks
  Surface area of papular areas in marker lesion (mm2)

CONTACTS AND LOCATIONS:
Overall Officials: Nevine H Kheir El Din, Prof., Study Director — Faculty of Dentistry-ASU
Locations (1):
- FUE, New Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Age, gender and the number of the participants
Supporting Information: Study Protocol, ICF
Time Frame: One year
Access Criteria: Accessibility for oral medicine researchers